CLINICAL TRIAL: NCT02070172
Title: A Comparison of Range of Motion During the Active and Passive Flexion-rotation Tests in Subjects Patients With Cervicogenic Headache
Brief Title: Active and Passive Cervical Flexion-rotation Tests
Status: Completed | Type: Observational
Sponsor: Des Moines University (Other)
Responsible Party: Principal Investigator, Shannon Petersen, Associate Professor, Doctor of Physical Therapy Program, Des Moines University
Other Study IDs: DMUSP2
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cervicogenic Headaches
Keywords: headache diagnosis; flexion rotation test; range of motion; upper cervical
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — This study compares observation of neck range of motion measures during the flexion rotation test (combining neck flexion with neck rotation) in two groups of subjects, one group has headaches and one groups is a healthy, asymptomatic group.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervicogenic Headache Group: This group of subjects is considered the symptomatic group. No intervention was provided in this study so there are no intervention groups.
- Healthy, Asymptomatic Group: Subjects in this group had no headache symptoms. Their neck motion was compared to subjects in the headache group. No intervention was provided to subjects in either group for this study.

SUMMARY:
Motion limitations have been previously reported in people with headaches originating from the neck/cervicogenic headaches. A test involving flexing and rotating the neck has been found useful to diagnose this type of headache. This observational study investigates this neck motion test when performed actively by the patient and passively by the examiner, then compares the results of motion attained.

ELIGIBILITY:
Inclusion Criteria:

* One-sided headaches
* Headaches caused by neck movement or sustained head positioning
* Neck, shoulder, or arm pain
* Intermittent headaches at least one headache per week for greater than 2 months
* Headaches of moderate intensity

Exclusion Criteria:

* A diagnosis of rheumatoid arthritis
* Current pregnancy
* International Headache Society criteria for other headache forms (such as tension or migraine)
* Cervical radiculopathy
* Treatment for headaches by a physical therapist, chiropractor, massage therapist, or osteopath in the past month
* Positive test for vertebral artery insufficiency or cranial-vertebral ligament instability

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: two groups of subjects were included; those with cervicogenic headaches and an asymptomatic group of healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion in degrees with the Flexion Rotation Test | Baseline only
  Two versions of this test were examined. A motion analysis system was used to measure degrees of motion. The test was done in two ways on each subject. Subjects sat in a chair, looked downward, then rotated their head/neck each direction. Subjects laid on their back while an examiner lifted their head, then rotated it each direction (same motion as described for the active test in the previous sentence).
  Within session reliability was also examined.

SECONDARY OUTCOMES:
Northwick park neck disability index | Baseline only
  This self-report questionnaire was completed by subjects prior to testing. It was not re-assessed as an outcome but rather used for baseline description of the subjects included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Petersen, PT, DScPT, Principal Investigator — Des Moines University
Locations (1):
- Des Moines University, Des Moines, Iowa, United States